CLINICAL TRIAL: NCT04429217
Title: Immediate vs Delayed Weight-bearing After Surgical Treatment of Malleolar Fractures: a Randomized Controlled Trial
Brief Title: A Study to Compare Two Different Managements After Ankle Surgery: Immediate and Delayed Weight-bearing.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORL-ORT-012
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Lateral Malleolus Fracture
Keywords: Ankle; surgical treatment; malleolar fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: clinical assessments will be assessed by an investigator blinded with respect to the rehabilitation regimen and all outcomes will be analysed by a statistician blinded to the moment when they were registered / administered (baseline or time points after randomization).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-A (Experimental): experimental post-operative rehabilitation intervention consisting in immediate weight-bearing
  Interventions: Other: immediate post-operative complete weight-bearing after surgery
- Arm-B (Active Comparator): control post-operative rehabilitation intervention consisting in delayed weight-bearing
  Interventions: Other: delayed weight-bearing for 6 weeks after surgery

INTERVENTIONS:
Other: immediate post-operative complete weight-bearing after surgery — Patients randomized to the experimental post-operative rehabilitation intervention will undergo to immediate complete weight-bearing starting immediately after surgery. Immediate complete weight-bearing consists in the possibility to undergo all the everyday activities without limiting weight-bearing and without the use of walking aids.
  During the rehabilitation period, patients will wear an ankle brace (VACOankle® OPED); this will ensure the safety of the early recovery phases, protecting from dangerous movements while allowing the mobilization in the healthy range of movement.
  Arms: Arm-A
Other: delayed weight-bearing for 6 weeks after surgery — Patients randomized to the control post-operative rehabilitation intervention will undergo to delayed weight-bearing starting at 6-weeks post-operatively. Delayed weight-bearing consists in the limitation of the weight-bearing to 20-30% of patient's total weight using crutches for the first 6 weeks after surgery.
  During the rehabilitation period, patients will wear an ankle brace (VACOankle® OPED).
  Arms: Arm-B

SUMMARY:
The investigators will compare two types of rehabilitation in patients who undergo a surgery for treatment of malleolar fractures: immediate complete weight-bearing and delayed weight-bearing.

The investigators want to evaluate if the immediate complete weight-bearing can improve and hasten the functional outcome of the ankle without increasing the risk of complications.

DETAILED DESCRIPTION:
The study population corresponds to the patients who may benefit from a post-operative rehabilitation protocol with immediate weight-bearing. Eligible lateral malleolar fractures are limited to Weber A and Weber B fractures, since they have a higher stability, after open reduction and internal fixation, compared to Weber C and Maisonneuve fractures. This higher stability gives the possibility to evaluate the benefit of the immediate weight-bearing protocol without safety concerns.

A power analysis was performed to estimate the required sample size to detect a significant difference in the OMAS score at 6 weeks between groups: the number of patients needed is 42 patients per group (84 patients overall) but, considering the risk of drop-outs, the investigators plan to enroll 20% more patients for a total of 100 patients.

The surgical operation will be carried out following the AO Foundation general and specific rules concerning the surgical treatment of malleolar fractures . In particular,an anatomical open reduction and internal fixation with one or two compression screws sustained by a neutralization third-tubular plate for simple fractures or a bridging third-tubular locking compression plate for multi-fragmentary fractures will be performed.

Postoperatively, patients who still meet the eligibility criteria will be randomized in 2 groups: immediate post-operative complete weight-bearing and complete weight-bearing delayed for 6 weeks.Immediate complete weight-bearing consists in the possibility to undergo all the everyday activities without limiting weight-bearing and without the use of walking aids (patients will wear an ankle brace, this will ensure the safety of the early recovery phases, protecting from dangerous movements while allowing the mobilization in the healthy range of movement). Delayed weight-bearing consists in the limitation of the weight-bearing to 20-30% of patient's total weight using crutches for the first 6 weeks after surgery (also patients of the control group will wear the ankle brace).

Subsequent follow-up visits are scheduled at 2, 6, 12 and 24 weeks after surgery. Patients with a fracture non-union radiologically confirmed at week 24 will be followed up until 48 weeks after surgery. Clinical assessments will be performed using subjective, objective and radiological evaluations. Safety will be monitored throughout the study.

Overall study duration will be 2 years and 6 months (2 years to reach the expected sample size and 6 months to complete the follow-up):

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults
* Age ranging from 18 to 70 years, included
* Signed Informed Consent
* Ankle fracture requiring surgical management classified as:1- Weber A fracture pattern (AO 44.A1, 44.A2, 44.A3) with or without association with a medial or posterior lesion/fracture or 2- Weber B fracture pattern (AO 44.B1, 44.B2, 44.B3) with or without association with a medial or posterior lesion/fracture
* Willingness and ability to participate in the trial

Exclusion Criteria:

* Weber C fracture pattern
* Bilateral fractures or fractures in other locations
* Maissoneauve associated lesion
* Body Mass Index < 18.5 and ≥ 30
* Metabolic diseases influencing fracture healing processes
* Medical comorbidities precluding operative intervention
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, general physical problem of the participant, etc.
* Inability or contraindications to undergo the investigated intervention
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2028-02-02 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
change from day 1 after surgery in subjective functional ankle recovery on the Olerud-Molander Ankle Score at week 6 | baseline and week 6
  Functional ankle recovery is measured using the Olerud-Molander Ankle Score (OMAS)- The OMAS is a validated, self-administered patient questionnaire designed to subjectively evaluate ankle function after fracture. The scale is an ordinal functional rating scale based on nine different items given different points.
  The total score is calculated as the sum of each rated item and range from 0 points (totally impaired function) to 100 points (completely unimpaired function). The OMAS questionnaire will be administered after surgery (visit 1, day 1) and at week 6 (visit 3).
  A negative change from the day of surgery to week 6 will indicate an improvement in OMAS score and, therefore, in functional ankle recovery.

SECONDARY OUTCOMES:
change in subjective functional ankle recovery on the Olerud-Molander Ankle Score during the first 24 weeks after surgery | baseline, week2, week 12 and week 24
  measured using the OMAS score at 2, 12 and 24 weeks postoperatively. measured using the Olerud-Molander Ankle Score (OMAS)- The OMAS is a validated, self-administered patient questionnaire designed to subjectively evaluate ankle function after fracture. The scale is an ordinal functional rating scale based on nine different items given different points.
  The total score is calculated as the sum of each rated item and range from 0 points (totally impaired function) to 100 points (completely unimpaired function). The OMAS questionnaire will be administered after surgery (visit 1, day 1) and at week 2 (visit 2), 12 (visit 4) and 24 (visit 5). A negative change from the day of surgery to week 2, 12 or 24 will indicate an improvement in OMAS score and, therefore, in functional ankle recovery.
Change form day of surgery in functional ankle disability on the Foot and Ankle Disability Index (FADI) during the first 24 weeks after surgery | baseline, 2, 6, 12 and 24 weeks
  measured using the Foot and Ankle Disability Index (FADI) at 2, 6, 12 and 24 weeks postoperatively.
  FADI is designed to assess functional limitations related to foot and ankle conditions. FADI consists of 4 pain-related and 22 activity-related items) for a total of 26.
  Each of the 22 activity-related items is scored on a 5-point Likert scale from 0 (unable to do) to 4 (no difficulty at all). The 4 pain-items are scored from 0 (none) to 4 (unbearable). The total FADI score is calculated as percentages, with 100% representing no ankle dysfunction.
  The FADI questionnaire will be administered after surgery (visit 1, day 1) and at week 2, (visit 2), 6 (visit 3), 12 (visit 4) and 24 (visit 5).
  A positive change from the day of surgery to week 2, 6, 12 or 24 will indicate an improvement in FADI score and, therefore, in functional ankle disability.
Change form baseline in pain on the Numerical Rating Scale (NRS) | baseline, 12 and 24 weeks
  measured by using a Numerical Rating Scale (NRS) at 12 and 24 weeks postoperatively.
  The pain NRS is a self-assessment scale in which patients rate their pain on an 11-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). The pain NRS will be administered after surgery (visit 1, day 1) and at 12 (visit 4) and 24 (visit 5).
  A negative change from the day of surgery to week 12 or 24 will indicate an improvement in pain NRS score and, therefore, in local pain.
Daily pain and function | 12 weeks
  monitored through mobile NRS application up to 12 weeks postoperatively. A new application suitable for the use with both Android and iOS running mobile phones was developed by our Institution (EOC- Ente Osedaliero Cantonale) , namely "EOC - EMApp". The application asks the patients two simple questions: to rate actual pain and function on a 0-10 NRS two times daily at random hours in the morning and the evening, as suggested by previous experiences. The following parameters will be calculated and compared between groups: average daily pain and function, mean value of pain and function for each week and for the entire period of assessment (12 weeks). If the patient does not have a smartphone, he/she will not be included it in this assessment group.
change in quality of life on the 36-Item Short Form Health Survey (SF-36 questionnaire). | baseline, 2, 6,12 and 24 weeks
  measured from the day of surgery (Day 1) to 2, 6, 12 and 24 weeks postoperatively by a using the SF-36 questionnaire.
  The SF-36 is a validated, self-administered questionnaire specifically designed for evaluating patient health-related quality of life. It comprises of 36 questions, relating to eight key areas of physical and psychological health, including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. The weighted-score of each area is transformed into a 0-100 scale, with lower scores indicating the more disability and higher scores the less disability.
  A negative change from the day of surgery to week 2, 6, 12 or 24 will indicate an improvement in SF-36 score and, therefore, in quality of life.
Return to previous daily activities on the Tegner activity level scale | week 12 and week 24
  evaluated by using the Tegner score at 12 and 24 weeks postoperatively. The Tegner activity level scale is a patient-administered rating system designed to provide a standardized method of grading work and sporting activities. It consists of a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury. The score varies from 0 that represents sick leave or disability pension because of ankle problems to 10 that corresponds to participation in national and international elite competitive sports.
  The Tegner activity level scale questionnaire will be administered at week 12 (visit 4) and 24 (visit 5).
  A positive change from score before injury to post-operative score will indicate an improvement in Tegner activity level scale score and, therefore, a higher level of activity and return to previous daily activity.
Objective ankle functional recovery | 6, 12, 24 weeks
  evaluated through gait analysis by using the OptoGait® at 6, 12, 24 weeks postoperatively.
  The OptoGait® is an avant-garde laser and video technology that permits to quantitatively measure through a sophisticated software the symmetry of the steps, the weight-bearing area, the time of foot-rest on the ground and other parameters. The change of each of this parameter will be evaluated at week 6 (visit 3), 12 (visit 4), 24 (visit 5) to assess the ankle functional recovery during the rehabilitation intervention.
Ankle joint flexibility | 6, 12, 24 weeks
  measured through the Ankle Range of Motion (ROM) assessed with a goniometer at 6, 12, 24 weeks postoperatively.
Objective activity level | 24 weeks
  Objective activity level will be continuously documented through a wrist activity tracker measuring daily walking distance up to 24 weeks. The patient will receive the tracker after the surgery and wear it for 24 weeks. The tracker, then, will be returned to the hospital during visit 5.
Radiological assessment | 24 weeks
  Standard X-ray assessment to determine healing, hardware fixation, fracture alignment, fracture reduction, implants mobilization will be performed at week 6 (visit 3), 12 (visit 4), 24 (visit 5). X-ray at 24 weeks will be done only in case of fracture non-union reported at the 12-weeks post-operatively.
Pain drug consumption | 24 weeks
  Pain drug consumption will be assessed by recording in a patient diary type and dosage of pain drugs, and reason for taking the drug from surgery (day 1, visit 1) up to 24 weeks (visit 5) postoperatively.
  Drug consumption will be quantified in milligrams of active principle taken per week and in number of days in which the patient required a pain drugs during the study period.
Patient satisfaction on the satisfaction Numerical Rating Scale (NRS scale) | day of surgery, week 6, 12 and 24
  Patient satisfaction will be documented by using 0-10 NRS administered at 6, 12, 24 weeks postoperatively. The satisfaction NRS is a self-assessment scale in which patients rate their satisfaction on an 11-point numerical scale from 0 (completely dissatisfied) to 10 (completely satisfied). The satisfaction NRS will be administered after surgery (visit 1, day 1) and at week 6 (visit 3), 12 (visit 4) and 24 (visit 5).
  A positive change from the day of surgery to week 6, 12 or 24 will indicate an improvement in satisfaction NRS score and, therefore, in patient satisfaction.

OTHER OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by the Clavien-Dindo classification. | from surgery up to 48 weeks
  The safety will be evaluated by documenting the incidence, nature and severity of all (serious) adverse events / post-operative complications that may in any way be related to the surgical procedure. In particular, wound complications, mal-union or non-union, fracture displacement, hardware failure requiring re-operations will be assessed.
  Incidence, nature and severity of all serious and adverse events / complications will be recorded. Severity will be assessed using the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Adrian Testa, MD, Principal Investigator — EOC
Locations (1):
- Ente Ospedaliero Cantonale, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No